CLINICAL TRIAL: NCT00607178
Title: Randomized, Single-Blind, Placebo-Controlled Study of Influenza Vaccine in Preventing Cardiovascular Events in Post-Myocardial Infarction Patients and in Those With Stable Angina Pectoris
Brief Title: The Efficacy of Influenza Vaccine in Reducing Cardiovascular Events in Patients With Coronary Artery Diseases
Acronym: IVCAD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Maryam Keshtkar-Jahromi, Infectious Diseases and Tropical Medicine Research Center, SBMU, Tehran, Iran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SBMU- 86-03-105-5433A; SMMC- 13861008A
Record Dates: First submitted 2008-01-10; First posted 2008-02-05 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2008-09

CONDITIONS: Coronary Artery Diseases; Myocardial Infarction; Stable Angina
Keywords: Influenza; Vaccine
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Angina, Stable; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Influenza vaccine (Experimental): Enrolled patients who are randomly assigned to receive influenza vaccine
  Interventions: Biological: influenza vaccine
- Placebo (Placebo Comparator): Enrolled patients who are randomly assigned to receive placebo of influenza vaccine
  Interventions: Biological: placebo for influenza vaccine

INTERVENTIONS:
Biological: influenza vaccine — Intramuscular injection of one 0.5-mL dose of influenza vaccine
  Other Names: 2006-2007 vaccination campaign of Influvac (SolvayPharma)
  Arms: Influenza vaccine
Biological: placebo for influenza vaccine — Intramuscular injection of one 0.5-mL dose of placebo for influenza vaccine
  Arms: Placebo

SUMMARY:
Influenza vaccine reduces the cardiovascular events in post-myocardial infarction (MI) patients and in those with stable angina (SA).

DETAILED DESCRIPTION:
A connection between infectious processes and atherosclerosis is repeatedly reported [1]. Acute respiratory infection was found to be associated with myocardial infarction (MI) [2,3] and a number of epidemiological studies found that mortality attributable to cardiovascular diseases is increased during influenza epidemics [4]. Naghavi et al [5] in a case-control study of patients with coronary artery disease (CAD) found that vaccination against influenza was negatively associated with the development of new MI during the same influenza season. While some clinical trials found influenza vaccine effective in secondary prevention of cardiovascular adverse events [6,7], a large trial [8] failed to approve such an efficacy. Furthermore, a recent review of published trials on the subject concluded that frailty selection bias and use of non-specific endpoints such as all cause mortality have led cohort studies to greatly exaggerate vaccine benefits and that the remaining evidence base is currently insufficient to indicate the magnitude of the mortality benefit of the vaccination program [9].

This study aims to assess the efficacy of vaccine in secondary prevention of cardiovascular events in MI and stable angina (SA) patients using specific endpoints including reliable quantitative tools.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of acute, evolving or recent MI (after recovered the acute phase) as defined by:

  1. Typical rise and gradual fall (troponin) or more rapid rise and fall (CK-MB) of biochemical markers of myocardial necrosis with at least one of the following:

     * Ischemic symptoms
     * Development of pathologic Qwaves on the ECG
     * ECG changes indicative of ischemia (ST segment elevation or depression); OR
     * Coronary artery intervention (e.g., coronary angioplasty).
  2. Pathologic findings of an acute MI [12]
* Patients with stable angina pectoris and documented coronary artery stenosis (angiography).

Exclusion Criteria:

* Any acute disease
* Chronic liver or kidney diseases
* Conditions accompanied by immunosuppression (like organ transplantation, HIV)
* Diagnosed malignancy
* Incubation with influenza vaccine within the past 5 years
* Any psychological disease that interferes with regular follow-up
* Congestive heart failure (Killip class IV)
* Unstable angina, and contradictions of vaccine incubation (like egg allergy).

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Cardiovascular death | 6 months

SECONDARY OUTCOMES:
Acute coronary syndrome (MI or unstable angina) | 6 months
Admission for Coronary Artery Disease | 6 months
Angina severity (Seattle Angina Questionnaire [10]) | 6 months
Coronary artery stenosis (modified Gensini score [11]) | 6 months
Coronary revascularization (artery bypass graft or percutaneous coronary intervention) | 6 months
Influenza infection | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Keshtkar-Jahromi, M.D.; M.P.H., Study Chair — Infectious Diseases and Tropical Medicine Research Center, Shaheed Beheshti Medical University, Tehran, Iran; Hossein Vakili, M.D., Principal Investigator — Cardiovascular Research Center, Shaheed Beheshti Medical University, Tehran, Iran; Ali Eskandari, MD, Principal Investigator — Shahid Beheshti University of Medical Sciences; Mohammad Rahnavardi, MD, Principal Investigator — Shahid Beheshti University of Medical Sciences; Sharareh Gholamin, MD, Principal Investigator — Shaheed Beheshti University (MC); Seyed Mostafa Razavi, MD, Principal Investigator — Shaheed Beheshti University (MC)
Locations (1):
- Shaheed Modarres Medical Center, Tehran, Tehran Province, Iran

REFERENCES:
- [Background] Gurfinkel E, Lernoud V. The role of infection and immunity in atherosclerosis. Expert Rev Cardiovasc Ther. 2006 Jan;4(1):131-7. doi: 10.1586/14779072.4.1.131. PMID 16375635
- [Background] Spodick DH, Flessas AP, Johnson MM. Association of acute respiratory symptoms with onset of acute myocardial infarction: prospective investigation of 150 consecutive patients and matched control patients. Am J Cardiol. 1984 Feb 1;53(4):481-2. doi: 10.1016/0002-9149(84)90016-x. PMID 6695777
- [Background] Bainton D, Jones GR, Hole D. Influenza and ischaemic heart disease--a possible trigger for acute myocardial infarction? Int J Epidemiol. 1978 Sep;7(3):231-9. doi: 10.1093/ije/7.3.231. PMID 721358
- [Background] Gurevich VS. Influenza, autoimmunity and atherogenesis. Autoimmun Rev. 2005 Feb;4(2):101-5. doi: 10.1016/j.autrev.2004.10.006. Epub 2004 Nov 20. PMID 15722256
- [Background] Naghavi M, Barlas Z, Siadaty S, Naguib S, Madjid M, Casscells W. Association of influenza vaccination and reduced risk of recurrent myocardial infarction. Circulation. 2000 Dec 19;102(25):3039-45. doi: 10.1161/01.cir.102.25.3039. PMID 11120692
- [Background] Gurfinkel EP, de la Fuente RL, Mendiz O, Mautner B. Influenza vaccine pilot study in acute coronary syndromes and planned percutaneous coronary interventions: the FLU Vaccination Acute Coronary Syndromes (FLUVACS) Study. Circulation. 2002 May 7;105(18):2143-7. doi: 10.1161/01.cir.0000016182.85461.f4. PMID 11994246
- [Background] Leon de la Fuente R, Gurfinkel EP, Toledo D, Mautner B; Grupo de Estudio FLUVACS. [Flu vaccination in patients with acute coronary syndromes: treatment benefit in prespecified subgroups]. Rev Esp Cardiol. 2003 Oct;56(10):949-54. doi: 10.1016/s0300-8932(03)76991-7. Spanish. PMID 14563288
- [Background] Jackson LA, Yu O, Heckbert SR, Psaty BM, Malais D, Barlow WE, Thompson WW; Vaccine Safety Datalink Study Group. Influenza vaccination is not associated with a reduction in the risk of recurrent coronary events. Am J Epidemiol. 2002 Oct 1;156(7):634-40. doi: 10.1093/aje/kwf073. PMID 12244032
- [Background] Simonsen L, Taylor RJ, Viboud C, Miller MA, Jackson LA. Mortality benefits of influenza vaccination in elderly people: an ongoing controversy. Lancet Infect Dis. 2007 Oct;7(10):658-66. doi: 10.1016/S1473-3099(07)70236-0. PMID 17897608
- [Background] Spertus JA, Winder JA, Dewhurst TA, Deyo RA, Prodzinski J, McDonell M, Fihn SD. Development and evaluation of the Seattle Angina Questionnaire: a new functional status measure for coronary artery disease. J Am Coll Cardiol. 1995 Feb;25(2):333-41. doi: 10.1016/0735-1097(94)00397-9. PMID 7829785
- [Background] Gensini GG. Coronary Angiography. Mount Kisco, NY: Futura Publishing Co; 1975.
- [Background] Alpert JS, Thygesen K, Antman E, Bassand JP. Myocardial infarction redefined--a consensus document of The Joint European Society of Cardiology/American College of Cardiology Committee for the redefinition of myocardial infarction. J Am Coll Cardiol. 2000 Sep;36(3):959-69. doi: 10.1016/s0735-1097(00)00804-4. PMID 10987628
- [Derived] Dehesh M, Gholamin S, Razavi SM, Eskandari A, Vakili H, Rahnavardi Azari M, Wang Y, Gough EK, Keshtkar-Jahromi M. Influenza Vaccination and Cardiovascular Outcomes in Patients with Coronary Artery Diseases: A Placebo-Controlled Randomized Study, IVCAD. Vaccines (Basel). 2025 Apr 27;13(5):472. doi: 10.3390/vaccines13050472. PMID 40432084